CLINICAL TRIAL: NCT01346969
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, WITHIN-SUBJECT CONTROLLED STUDY TO EVALUATE EFFICACY AND SAFETY OF VARIOUS DOSES AND REGIMENS OF EXC 001 FOR THE AMELIORATION OF SCARRING FOLLOWING REVISION OF SCARS FROM PRIOR BREAST SURGERY IN ADULT SUBJECTS (LEGACY EXCALIARD PROTOCOL # EXC 001-204)
Brief Title: Safety and Efficacy Study of EXC 001 to Improve the Appearance of Scars From Prior Breast Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: EXC 001-204; B5301004 (Other: Alias Study Number)
Record Dates: First submitted 2011-05-01; First posted 2011-05-04 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Reduction in Hypertrophic Skin Scarring
Keywords: Skin scarring; cicatrix; breast scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator)
  Interventions: Drug: EXC 001
- Group 2 (Placebo Comparator)
  Interventions: Drug: EXC 001
- Group 3 (Placebo Comparator)
  Interventions: Drug: EXC 001
- Group 4 (Placebo Comparator)
  Interventions: Drug: EXC 001

INTERVENTIONS:
Drug: EXC 001 — Single-dose administered by injection four different times
  Arms: Group 1
Drug: EXC 001 — Single reduced dose compared to Group 1 administered by injection at the same four time periods as Group 1
  Arms: Group 2
Drug: EXC 001 — Single reduced dose compared to Groups 1 and 2 administered by injection at the same four time periods as Groups 1 and 2
  Arms: Group 3
Drug: EXC 001 — Same sinlge dose as Group 1 administered by injection at the same four time periods as Groups 1, 2, and 3
  Arms: Group 4

SUMMARY:
The study will investigate the efficacy of various doses and regimens of EXC 001 in reducing skin scarring in subjects undergoing revision of scars from prior surgery. The study will also evaluate the safety and tolerability of EXC 001 and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have previous had breast surgery resulting in unacceptable scars.
* Subject has chosen to have breast scars revised.
* Subject must not be pregnant or lactating.

Exclusion Criteria:

* Currently pregnant or pregnant during the 6 months, prior to inclusion in the study or lactating.
* Participation in another clinical trial within 30 days prior to the start of the study.
* Any other condition or prior therapy, which, in the opinion of the PI, would make the subject unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2012-04-16 (Actual); Study Completion 2012-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Skin Deep Laser Medical Spa, Pasadena, California
  - Bright Health Physicans Plastic Surgery and Aesthetic Medicine, Whittier, California
  - Altus Research, Lake Worth, Florida
  - Bayside Ambulatory Center, Miami, Florida
  - Aesthetic Plastic Surgery Miami, Miami, Florida
  - Body Aesthetic Plastic Surgery, St Louis, Missouri
  - New Jersey Plastic Surgery, Montclair, New Jersey
  - Mark L. Jewell,MD Surgery Center, Eugene, Oregon
  - Connall Consmetic Surgery, Tualatin, Oregon
  - Endeavor Clinical Trials,P.A., San Antonio, Texas
  - Texas Plastic Surgery, San Antonio, Texas
  - BAXTER Plastic Surgery, Mountlake Terrace, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=EXC001-204&StudyName=Safety%20and%20Efficacy%20Study%20of%20EXC%20001%20to%20Improve%20the%20Appearance%20of%20Scars%20From%20Prior%20Breast%20Surgery

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who previously had breast surgery resulting in unacceptable bilateral scars and had chosen to have the breast scars revised were recruited in this study.
Groups:
- EXC 001 (PF-06473871) 5 mg/cm: Participants received 4 intradermal injections of EXC 001 (PF- 06473871) at dose of 5 milligram per linear centimeter (mg/cm) at Week 2, 5, 8 and 11 to a 5 centimeter (cm) section of both sides of the revised scar on 1 breast and 3 intradermal injections of EXC 001 at dose of 5 mg/cm at Week 2, 5, 8 and then 1 intradermal injections of placebo matched to EXC 001 (PF- 06473871) at Week 11 to 5 cm section of both sides of the revised scar on another breast.
- EXC 001 (PF-06473871) 2 mg/cm and Placebo: Participants received 4 intradermal injections of EXC 001 (PF- 06473871) at dose of 2 mg/cm at Week 2, 5, 8 and 11 to a 5 cm section of both sides of the revised scar on 1 breast and 4 intradermal injections of placebo matched to EXC 001 (PF- 06473871) at Week 2, 5, 8 and 11 to 5 cm section of both sides of the revised scar on another breast.
- EXC 001 (PF-06473871) 0.8 mg/cm and Placebo: Participants received 4 intradermal injections of EXC 001 (PF- 06473871) at dose of 0.8 mg/cm at Week 2, 5, 8 and 11 to a 5 cm section of both sides of the revised scar on 1 breast and 4 intradermal injections of placebo matched to EXC 001 (PF- 06473871) at Week 2, 5, 8 and 11 to 5 cm section of both sides of the revised scar on another breast.
- EXC 001 (PF-06473871) 5 mg/cm and Placebo: Participants received 4 intradermal injections of EXC 001 (PF- 06473871) at dose of 5 mg/cm at Week 2, 5, 8 and 11 to a 5 cm section of both sides of the revised scar on 1 breast and 4 intradermal injections of placebo matched to EXC 001 (PF- 06473871) at Week 2, 5, 8 and 11 to 5 cm section of both sides of the revised scar on another breast.
Period: Overall Study
Arm/Group | EXC 001 (PF-06473871) 5 mg/cm | EXC 001 (PF-06473871) 2 mg/cm and Placebo | EXC 001 (PF-06473871) 0.8 mg/cm and Placebo | EXC 001 (PF-06473871) 5 mg/cm and Placebo
Started | 28 | 14 | 13 | 13
Safety Population | 27 | 14 | 13 | 13
Completed | 26 | 14 | 10 | 12
Not Completed | 2 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Randomized but not treated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population was defined as all participants that have missed no more than 1 dose of study medication.
Groups:
- EXC 001 (PF-06473871) 5 mg/cm: Participants received 4 intradermal injections of EXC 001 (PF- 06473871) at dose of 5 mg/cm at Week 2, 5, 8 and 11 to a 5 cm section of both sides of the revised scar on 1 breast and 3 intradermal injections of EXC 001 at dose of 5 mg/cm at Week 2, 5, 8 and then 1 intradermal injections of placebo matched to EXC 001 (PF- 06473871) at Week 11 to 5 cm section of both sides of the revised scar on another breast.
- Total: Total of all reporting groups
Arm/Group | EXC 001 (PF-06473871) 5 mg/cm | EXC 001 (PF-06473871) 2 mg/cm and Placebo | EXC 001 (PF-06473871) 0.8 mg/cm and Placebo | EXC 001 (PF-06473871) 5 mg/cm and Placebo | Total
Number analyzed (Participants) | 26 | 14 | 11 | 12 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (10.9) | 43.2 (7.16) | 40.1 (13.29) | 38.4 (8.22) | 39.9 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 14 | 11 | 11 | 62
  Male | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Physician Observer Scar Assessment Score at Week 24
Description: Physician assessment of scar was done using a valid published 10-point rating scale. Physician rated vascularity, pigmentation, thickness, relief, pliability, surface area and overall opinion for scar on a score of 1 = normal skin to 10 = worst scar imaginable, where lower scores indicated better outcome. Composite score was the sum of all the scores, except the overall opinion score, and range from 6 (best score) to 60 (worst score), where lower scores indicated better outcome. Within participant treatment difference was assessed between the treatment regimens each participant received.
Time Frame: Week 24
Population: Analysis population included all participants who missed not more than 1 dose of study drug, had physician observer scar assessment score at all specified time-points. Here 'N' (Overall Number of Participants Analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXC 001 (PF-06473871) 5 mg/cm | EXC 001 (PF-06473871) 2 mg/cm and Placebo | EXC 001 (PF-06473871) 0.8 mg/cm and Placebo | EXC 001 (PF-06473871) 5 mg/cm and Placebo
Number analyzed (Participants) | 26 | 14 | 10 | 12
units on a scale
  Overall Opinion | 0.0 (1.92) | -0.5 (2.31) | 0.8 (1.87) | -0.3 (1.97)
  Vascularity | 0.0 (1.70) | -0.6 (1.91) | 0.9 (1.52) | -0.2 (1.64)
  Pigmentation | -0.3 (1.41) | -0.4 (2.10) | 0.7 (1.42) | -0.3 (1.36)
  Thickness | 0.2 (2.41) | -0.6 (2.38) | 0.8 (2.04) | -0.2 (1.90)
  Relief | 0.0 (2.24) | -0.4 (1.95) | 0.7 (2.36) | -0.2 (1.90)
  Pliability | 0.2 (1.99) | -0.6 (2.27) | 0.6 (1.71) | -0.4 (1.62)
  Surface Area | 0.1 (1.75) | -0.4 (2.85) | 0.6 (1.90) | -0.1 (2.15)
  Composite Score | 0.2 (10.53) | -3.1 (12.60) | 4.3 (9.76) | -1.3 (8.67)
Statistical Analysis 1: Comparison: EXC 001 (PF-06473871) 5 mg/cm; Overall Opinion: Intraparticipant analysis; Test type: Other — LS Mean, SE, 95% confidence interval, and p-value were derived from MMRM model that includes fixed factors for treatment, pooled site, scheduled visit, an interaction for treatment by scheduled visit, and a covariate for Fitzpatrick category; p = 1.000, Mixed Models Analysis; LS Mean = 0.0, 95% CI 2-sided [-0.8 to 0.8], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: EXC 001 (PF-06473871) 5 mg/cm; Vascularity: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 1.000, Mixed Models Analysis; LS Mean = 0.0, 95% CI 2-sided [-0.7 to 0.7], Standard Error of Mean 0.37
Statistical Analysis 3: Comparison: EXC 001 (PF-06473871) 5 mg/cm; Pigmentation: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.391, Mixed Models Analysis; LS Mean = -0.3, 95% CI 2-sided [-1.0 to 0.4], Standard Error of Mean 0.36
Statistical Analysis 4: Comparison: EXC 001 (PF-06473871) 5 mg/cm; Thickness: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.696, Mixed Models Analysis; LS Mean = 0.2, 95% CI 2-sided [-0.6 to 0.9], Standard Error of Mean 0.39
Statistical Analysis 5: Comparison: EXC 001 (PF-06473871) 5 mg/cm; Relief: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.921, Mixed Models Analysis; LS Mean = 0.0, 95% CI 2-sided [-0.7 to 0.8], Standard Error of Mean 0.39
Statistical Analysis 6: Comparison: EXC 001 (PF-06473871) 5 mg/cm; Pliability: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.693, Mixed Models Analysis; LS Mean = 0.2, 95% CI 2-sided [-0.6 to 0.9], Standard Error of Mean 0.39
Statistical Analysis 7: Comparison: EXC 001 (PF-06473871) 5 mg/cm; Surface Area: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.770, Mixed Models Analysis; LS Mean = 0.1, 95% CI 2-sided [-0.7 to 0.9], Standard Error of Mean 0.39
Statistical Analysis 8: Comparison: EXC 001 (PF-06473871) 5 mg/cm; Composite Score: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.938, Mixed Models Analysis; LS Mean = 0.2, 95% CI 2-sided [-3.7 to 4.0], Standard Error of Mean 1.98
Statistical Analysis 9: Comparison: EXC 001 (PF-06473871) 2 mg/cm and Placebo; Overall Opinion: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.340, Mixed Models Analysis; LS Mean = -0.5, 95% CI 2-sided [-1.5 to 0.5], Standard Error of Mean 0.52
Statistical Analysis 10: Comparison: EXC 001 (PF-06473871) 2 mg/cm and Placebo; Vascularity: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.258, Mixed Models Analysis; LS Mean = -0.6, 95% CI 2-sided [-1.6 to 0.4], Standard Error of Mean 0.50
Statistical Analysis 11: Comparison: EXC 001 (PF-06473871) 2 mg/cm and Placebo; Pigmentation: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.381, Mixed Models Analysis; LS Mean = -0.4, 95% CI 2-sided [-1.4 to 0.5], Standard Error of Mean 0.49
Statistical Analysis 12: Comparison: EXC 001 (PF-06473871) 2 mg/cm and Placebo; Thickness: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.287, Mixed Models Analysis; LS Mean = -0.6, 95% CI 2-sided [-1.6 to 0.5], Standard Error of Mean 0.54
Statistical Analysis 13: Comparison: EXC 001 (PF-06473871) 2 mg/cm and Placebo; Relief: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.420, Mixed Models Analysis; LS Mean = -0.4, 95% CI 2-sided [-1.5 to 0.6], Standard Error of Mean 0.53
Statistical Analysis 14: Comparison: EXC 001 (PF-06473871) 2 mg/cm and Placebo; Pliability: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.227, Mixed Models Analysis; LS Mean = -0.6, 95% CI 2-sided [-1.7 to 0.4], Standard Error of Mean 0.53
Statistical Analysis 15: Comparison: EXC 001 (PF-06473871) 2 mg/cm and Placebo; Surface Area: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.427, Mixed Models Analysis; LS Mean = -0.4, 95% CI 2-sided [-1.5 to 0.6], Standard Error of Mean 0.54
Statistical Analysis 16: Comparison: EXC 001 (PF-06473871) 2 mg/cm and Placebo; Composite Score: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.256, Mixed Models Analysis; LS Mean = -3.1, 95% CI 2-sided [-8.4 to 2.2], Standard Error of Mean 2.70
Statistical Analysis 17: Comparison: EXC 001 (PF-06473871) 0.8 mg/cm and Placebo; Overall Opinion: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.198, Mixed Models Analysis; LS Mean = 0.8, 95% CI 2-sided [-0.4 to 2.0], Standard Error of Mean 0.62
Statistical Analysis 18: Comparison: EXC 001 (PF-06473871) 0.8 mg/cm and Placebo; Vascularity: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.132, Mixed Models Analysis; LS Mean = 0.9, 95% CI 2-sided [-0.3 to 2.1], Standard Error of Mean 0.60
Statistical Analysis 19: Comparison: EXC 001 (PF-06473871) 0.8 mg/cm and Placebo; Pigmentation: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.227, Mixed Models Analysis; LS Mean = 0.7, 95% CI 2-sided [-0.4 to 1.8], Standard Error of Mean 0.58
Statistical Analysis 20: Comparison: EXC 001 (PF-06473871) 0.8 mg/cm and Placebo; Thickness: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.208, Mixed Models Analysis; LS Mean = 0.8, 95% CI 2-sided [-0.4 to 2.0], Standard Error of Mean 0.63
Statistical Analysis 21: Comparison: EXC 001 (PF-06473871) 0.8 mg/cm and Placebo; Relief: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.265, Mixed Models Analysis; LS Mean = 0.7, 95% CI 2-sided [-0.5 to 1.9], Standard Error of Mean 0.63
Statistical Analysis 22: Comparison: EXC 001 (PF-06473871) 0.8 mg/cm and Placebo; Pliability: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.340, Mixed Models Analysis; LS Mean = 0.6, 95% CI 2-sided [-0.6 to 1.8], Standard Error of Mean 0.63
Statistical Analysis 23: Comparison: EXC 001 (PF-06473871) 0.8 mg/cm and Placebo; Surface Area: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.347, Mixed Models Analysis; LS Mean = 0.6, 95% CI 2-sided [-0.7 to 1.9], Standard Error of Mean 0.64
Statistical Analysis 24: Comparison: EXC 001 (PF-06473871) 0.8 mg/cm and Placebo; Composite Score: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.179, Mixed Models Analysis; LS Mean = 4.3, 95% CI 2-sided [-2.0 to 10.6], Standard Error of Mean 3.19
Statistical Analysis 25: Comparison: EXC 001 (PF-06473871) 5 mg/cm and Placebo; Overall Opinion: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.556, Mixed Models Analysis; Least Square (LS) Mean = -0.3, 95% CI 2-sided [-1.4 to 0.8], Standard Error of Mean 0.57
Statistical Analysis 26: Comparison: EXC 001 (PF-06473871) 5 mg/cm and Placebo; Vascularity: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.760, Mixed Models Analysis; LS Mean = -0.2, 95% CI 2-sided [-1.2 to 0.9], Standard Error of Mean 0.54
Statistical Analysis 27: Comparison: EXC 001 (PF-06473871) 5 mg/cm and Placebo; Pigmentation: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.636, Mixed Models Analysis; LS Mean = -0.3, 95% CI 2-sided [-1.3 to 0.8], Standard Error of Mean 0.53
Statistical Analysis 28: Comparison: EXC 001 (PF-06473871) 5 mg/cm and Placebo; Thickness: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.774, Mixed Models Analysis; LS Mean = -0.2, 95% CI 2-sided [-1.3 to 1.0], Standard Error of Mean 0.58
Statistical Analysis 29: Comparison: EXC 001 (PF-06473871) 5 mg/cm and Placebo; Relief: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.771, Mixed Models Analysis; LS Mean = -0.2, 95% CI 2-sided [-1.3 to 1.0], Standard Error of Mean 0.57
Statistical Analysis 30: Comparison: EXC 001 (PF-06473871) 5 mg/cm and Placebo; Pliability: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.468, Mixed Models Analysis; LS Mean = -0.4, 95% CI 2-sided [-1.5 to 0.7], Standard Error of Mean 0.57
Statistical Analysis 31: Comparison: EXC 001 (PF-06473871) 5 mg/cm and Placebo; Surface Area: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.886, Mixed Models Analysis; LS Mean = -0.1, 95% CI 2-sided [-1.2 to 1.1], Standard Error of Mean 0.58
Statistical Analysis 32: Comparison: EXC 001 (PF-06473871) 5 mg/cm and Placebo; Composite Score: Intraparticipant analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.668, Mixed Models Analysis; LS Mean = -1.3, 95% CI 2-sided [-7.0 to 4.5], Standard Error of Mean 2.91

2. Secondary Outcome: Physician Observer Scar Assessment Score
Description: Physician observer scar assessment score was done using a valid published 10-point rating scale. Physician rated vascularity, pigmentation, thickness, relief, pliability, surface area and overall opinion for a scar on a score of 1 = normal skin to 10 = worst scar imaginable, where lower scores indicated better outcome. Composite score was the sum of all the scores except the overall opinion score and range from 6 (best score) to 60 (worst score), where lower scores indicated better outcome. Within participant treatment difference was assessed between the treatment regimens each participant received.
Time Frame: Week 11, 18
Population: Analysis population included all participants who missed not more than 1 dose of study drug, had physician observer scar assessment score at all specified time-points. Here 'number analyzed' signifies those participants who were evaluable for this measure at specified time point for each group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXC 001 (PF-06473871) 5 mg/cm | EXC 001 (PF-06473871) 2 mg/cm and Placebo | EXC 001 (PF-06473871) 0.8 mg/cm and Placebo | EXC 001 (PF-06473871) 5 mg/cm and Placebo
Number analyzed (Participants) | 26 | 14 | 11 | 12
units on a scale
  Week 11, Overall Opinion: number analyzed (Participants) | 26 | 12 | 11 | 12
  Week 11, Overall Opinion | -0.3 (2.27) | -0.6 (2.07) | 0.2 (2.04) | 0.3 (1.54)
  Week 11, Vascularity: number analyzed (Participants) | 26 | 12 | 11 | 12
  Week 11, Vascularity | 0.0 (2.12) | -0.2 (1.70) | 0.1 (1.38) | 0.0 (1.21)
  Week 11, Pigmentation: number analyzed (Participants) | 26 | 12 | 11 | 12
  Week 11, Pigmentation | -0.5 (1.88) | -0.1 (1.78) | 0.4 (1.50) | 0.0 (1.54)
  Week 11, Thickness: number analyzed (Participants) | 26 | 12 | 11 | 12
  Week 11, Thickness | -0.4 (2.18) | -0.1 (2.15) | 0.2 (1.99) | -0.2 (1.85)
  Week 11, Relief: number analyzed (Participants) | 26 | 12 | 11 | 12
  Week 11, Relief | -0.4 (2.00) | -0.3 (2.05) | 0.0 (2.28) | 0.0 (2.26)
  Week 11, Pliability: number analyzed (Participants) | 26 | 12 | 11 | 12
  Week 11, Pliability | -0.4 (2.40) | -0.2 (2.29) | -0.2 (2.27) | -0.3 (1.76)
  Week 11, Surface Area: number analyzed (Participants) | 26 | 12 | 11 | 12
  Week 11, Surface Area | -0.4 (2.14) | -0.3 (2.27) | 0.1 (1.04) | 0.3 (1.82)
  Week 11, Composite Score: number analyzed (Participants) | 26 | 12 | 11 | 12
  Week 11, Composite Score | -2.1 (11.46) | -1.1 (11.19) | 0.5 (9.75) | -0.2 (8.57)
  Week 18, Overall Opinion: number analyzed (Participants) | 26 | 14 | 11 | 11
  Week 18, Overall Opinion | 0.1 (2.07) | -0.7 (2.43) | 0.3 (2.05) | 0.4 (2.25)
  Week 18, Vascularity: number analyzed (Participants) | 26 | 14 | 11 | 11
  Week 18, Vascularity | 0.3 (1.51) | -0.6 (2.24) | -0.1 (1.97) | 0.5 (1.57)
  Week 18, Pigmentation: number analyzed (Participants) | 26 | 14 | 11 | 11
  Week 18, Pigmentation | -0.2 (1.49) | -0.6 (2.34) | 0.3 (1.56) | 0.0 (1.79)
  Week 18, Thickness: number analyzed (Participants) | 26 | 14 | 11 | 11
  Week 18, Thickness | -0.1 (2.24) | -0.4 (2.28) | 0.5 (1.97) | 0.6 (2.29)
  Week 18, Relief: number analyzed (Participants) | 26 | 14 | 11 | 11
  Week 18, Relief | 0.2 (2.41) | -0.3 (2.49) | 0.5 (1.86) | 0.5 (2.21)
  Week 18, Pliability: number analyzed (Participants) | 26 | 14 | 11 | 11
  Week 18, Pliability | 0.2 (2.19) | -0.7 (2.52) | 0.5 (1.21) | 0.7 (2.24)
  Week 18, Surface Area: number analyzed (Participants) | 26 | 14 | 11 | 11
  Week 18, Surface Area | -0.1 (2.28) | -0.4 (2.50) | 0.4 (1.75) | 0.2 (2.40)
  Week 18, Composite Score: number analyzed (Participants) | 26 | 14 | 11 | 11
  Week 18, Composite Score | 0.4 (10.45) | -3.1 (13.44) | 2.1 (9.45) | 2.5 (11.21)

3. Secondary Outcome: Expert Panel Scar Assessment Score
Description: Scar assessment by an expert panel was done on blinded photographs using 100 millimeter (mm) visual analog scale (VAS) where a score of 0 = best possible scar and a score of 100 = worst possible scar, where lower scores indicated better outcome. The rater first marked a rating for the "worse" scar and then rated the other scar. The difference between these two ratings was the "improvement of scar severity." If there was no difference, the expert could check a box to indicate that determination. This method provided information on the absolute severity of the scars as well as the differences between the two scars in the pair.
Time Frame: Week 11, 18, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXC 001 (PF-06473871) 5 mg/cm | EXC 001 (PF-06473871) 2 mg/cm and Placebo | EXC 001 (PF-06473871) 0.8 mg/cm and Placebo | EXC 001 (PF-06473871) 5 mg/cm and Placebo
Number analyzed (Participants) | 26 | 14 | 11 | 12
units on a scale
  Week 11: number analyzed (Participants) | 26 | 13 | 11 | 12
  Week 11 | 2.0 (14.67) | 0.4 (15.89) | 3.7 (13.18) | -4.1 (13.71)
  Week 18 | 2.2 (14.70) | -2.7 (13.54) | 9.5 (14.28) | -2.1 (15.94)
  Week 24: number analyzed (Participants) | 26 | 14 | 10 | 12
  Week 24 | 4.1 (15.94) | -2.5 (17.78) | 6.5 (15.38) | -1.5 (15.43)

4. Secondary Outcome: Subject Observer Scar Assessment Score
Description: Participants rated pain, itching, color, stiffness, thickness, irregularity, and overall opinion of scar on 10-point scale. For pain and itching associated with scar: range = 1 (no, not at all) to 10 (yes, worst imaginable) and for other parameters associated with scar compared to normal skin: range = 1 (no, same as normal skin) to 10 (yes, very different). Composite score = sum of all scores except overall opinion and range 6 (best) to 60 (worst). Scar appearance composite score = sum of all scores except overall opinion, pain and itching, range 4 (best) to 40 (worst). Within participant treatment difference was assessed between the treatment regimens each participant received. A lower score indicated a better outcome.
Time Frame: Week 24
Population: Analysis population included all participants who missed not more than 1 dose of study drug, had physician observer scar assessment score at all specified time-points. Here 'N' (Overall Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXC 001 (PF-06473871) 5 mg/cm | EXC 001 (PF-06473871) 2 mg/cm and Placebo | EXC 001 (PF-06473871) 0.8 mg/cm and Placebo | EXC 001 (PF-06473871) 5 mg/cm and Placebo
Number analyzed (Participants) | 26 | 14 | 10 | 12
units on a scale
  Overall Opinion | -0.1 (2.47) | 0.0 (2.22) | 1.2 (2.35) | -0.2 (2.55)
  Pain | -0.2 (2.25) | 0.2 (0.89) | 0.3 (0.95) | -0.1 (0.51)
  Itching | 0.0 (1.11) | 0.1 (0.86) | 0.3 (0.95) | -0.3 (0.65)
  Color | -0.5 (1.58) | -0.1 (1.82) | 0.6 (1.17) | 0.3 (2.05)
  Stiffness | -0.4 (1.68) | 0.1 (2.06) | 0.4 (2.22) | -0.1 (3.00)
  Thickness | -0.2 (2.22) | 0.0 (1.36) | 0.7 (2.41) | 0.2 (3.19)
  Irregular | -0.3 (1.96) | -0.1 (1.96) | 0.7 (2.58) | 0.0 (3.05)
  Composite Score | -1.7 (9.03) | 0.2 (6.80) | 3.0 (8.52) | -0.1 (11.34)
  Scar Appearance Composite Score | -1.5 (6.77) | -0.1 (6.44) | 2.4 (7.68) | 0.3 (10.71)

5. Secondary Outcome: Number of Participants With Physician Photonumeric Guide Scar Assessment Score
Description: Physician rated severity of each scar using a photonumeric guide on a scale range from 1 to 5 (where 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe). Number of participants with different ratings of scar severity were reported. Same participant was reported twice, once for each breast's scar (dosing for 1 breast = 4 times EXC 001 and for other breast = 3 times).
Time Frame: Week 24
Population: Analysis population included all participants who missed not more than 1 dose of study drug, had physician observer scar assessment score at all specified time-points. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | EXC 001 (PF-06473871) 5 mg/cm | EXC 001 (PF-06473871) 2 mg/cm and Placebo | EXC 001 (PF-06473871) 0.8 mg/cm and Placebo | EXC 001 (PF-06473871) 5 mg/cm and Placebo
Number analyzed (Participants) | 26 | 14 | 10 | 12
Participants
  4 times EXC 001, minimal | 10 | 4 | 1 | 0
  4 times EXC 001, mild | 6 | 3 | 5 | 7
  4 times EXC 001, moderate | 3 | 3 | 3 | 1
  4 times EXC 001, severe | 6 | 3 | 0 | 2
  4 times EXC 001, very severe | 1 | 1 | 1 | 2
  3 times EXC 001/Placebo, minimal | 7 | 2 | 6 | 4
  3 times EXC 001/Placebo, mild | 13 | 5 | 1 | 0
  3 times EXC 001/Placebo, moderate | 2 | 2 | 1 | 3
  3 times EXC 001/Placebo, severe | 3 | 4 | 2 | 4
  3 times EXC 001/Placebo, very severe | 1 | 1 | 0 | 1

6. Secondary Outcome: Number of Participants With Participant Photonumeric Guide Scar Assessment Score
Description: Participants rated severity of each scar using a photonumeric guide on a scale range from 1 to 5 (where 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe). Number of participants with different ratings of scar severity were reported. Same participant was reported twice, once for each breast's scar (dosing for 1 breast = 4 times EXC 001 and for other breast = 3 times).
Time Frame: Week 24
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | EXC 001 (PF-06473871) 5 mg/cm | EXC 001 (PF-06473871) 2 mg/cm and Placebo | EXC 001 (PF-06473871) 0.8 mg/cm and Placebo | EXC 001 (PF-06473871) 5 mg/cm and Placebo
Number analyzed (Participants) | 26 | 13 | 10 | 12
Participants
  4 times EXC 001, minimal | 8 | 1 | 1 | 1
  4 times EXC 001, mild | 8 | 1 | 4 | 4
  4 times EXC 001, moderate | 2 | 4 | 3 | 4
  4 times EXC 001, severe | 7 | 5 | 1 | 2
  4 times EXC 001, very severe | 1 | 2 | 1 | 1
  3 times EXC 001/Placebo, minimal | 4 | 1 | 4 | 2
  3 times EXC 001/Placebo, mild | 13 | 3 | 2 | 3
  3 times EXC 001/Placebo, moderate | 4 | 4 | 1 | 2
  3 times EXC 001/Placebo, severe | 4 | 3 | 1 | 4
  3 times EXC 001/Placebo, very severe | 1 | 2 | 2 | 1

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 24
Arm/Group | EXC 001 (PF-06473871) 5 mg/cm | EXC 001 (PF-06473871) 2 mg/cm and Placebo | EXC 001 (PF-06473871) 0.8 mg/cm and Placebo | EXC 001 (PF-06473871) 5 mg/cm and Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/14 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 13/27 | 2/14 | 2/13 | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EXC 001 (PF-06473871) 5 mg/cm (N=27) | EXC 001 (PF-06473871) 2 mg/cm and Placebo (N=14) | EXC 001 (PF-06473871) 0.8 mg/cm and Placebo (N=13) | EXC 001 (PF-06473871) 5 mg/cm and Placebo (N=13)
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 1 | 0 | 0
Lyme disease (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Application site rash (General disorders) | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1
Breast induration (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.